CLINICAL TRIAL: NCT07302438
Title: Comparative Evaluation of Calcium Silicate-doped Treated Dentin Matrix and Mineral Trioxide Aggregate as Miniature Pulpotomy Biomaterials in Deep Carious Lesions: a Parallel, Double-blind, Randomised Clinical Trial
Brief Title: Comparative Evaluation of Calcium Silicate-doped Treated Dentin Matrix and Mineral Trioxide Aggregate as Miniature Pulpotomy Biomaterials in Deep Carious Lesions
Acronym: hTDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ganesh Jadhav, Associate Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/Pharmac/2024/1|04; CTRI/2025/04/084767 (Other: Clinical Trial Registry of India)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Reversible Pulpitis; Deep Carious Lesions
Keywords: Human treated dentin matrix; Mineral Trioxide Aggregate; Calcium silicate
MeSH Terms: interventions — mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care arm: (Control group) Mineral Trioxide Aggregate (MTA) for miniature pulpotomy (Experimental): Mineral Trioxide Aggregate (MTA) for miniature pulpotomy (MTA MP). MTA serves as a standard of care intervention
  Interventions: Procedure: Mineral Trioxide Aggregate (MTA) for Miniature Pulpotomy
- Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP). (Experimental): Procedure/Surgery: Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP).
  Description: Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP).
  Interventions: Procedure: Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP).

INTERVENTIONS:
Procedure: Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP). — Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP).
  Arms: Calcium Silicate doped treated dentin matrix for miniature pulpotomy (CaSi+hTDM MP).
Procedure: Mineral Trioxide Aggregate (MTA) for Miniature Pulpotomy — Mineral Trioxide Aggregate (MTA) for miniature pulpotomy. MTA serves as standard of care.
  Arms: Standard of Care arm: (Control group) Mineral Trioxide Aggregate (MTA) for miniature pulpotomy

SUMMARY:
AIM:

To compare the efficacy of a Novel calcium silicate doped treated dentin matrix and Mineral Trioxide aggregate as biomaterials for miniature pulpotomy.

OBJECTIVES:

Primary objective:

To evaluate the efficacy of calcium silicate-doped human-treated dentin matrix (CaSi+hTDM) compared to Mineral Trioxide Aggregate (MTA) in maintaining pulp vitality using cold testing following Miniature Pulpotomy (MP) in deep and extremely deep carious lesions with reversible pulpitis in 14- to 35-year-old patients reporting to Department of Dentistry, AIIMS Nagpur.

Secondary objectives:

1. To evaluate patient-reported outcomes such as pain, swelling, sinus tract etc. post-operatively.
2. To determine the clinical success rates of both materials by assessing the Periapical index of healing over a 6 months follow-up period.

NULL HYPOTHESIS:

The null hypothesis (H0) is that there is no difference between CaSi+hTDM and MTA in maintaining pulp vitality when used as a Miniature Pulpotomy (MP) biomaterial in carious lesions.

DETAILED DESCRIPTION:
1 INTRODUCTION The loss of tooth structure significantly affects the quality of life for patients. This loss occurs due to decay and other non-carious causes. The resulting inadequate aesthetics and impaired function affects even the psychological wellbeing of the patient. Conventional root canal therapy alongside a quality coronal restoration is widely regarded as the standard treatment for this issue. Yet, traditional treatment approaches consistently present challenges such as significant periradicular dentin loss and the risk of reinfection resulting from a compromised coronal seal. Ideally reestablishment of the lost tissue to their pre-disease level should be the goal of these treatment strategies. Regeneration of the dentin-pulp complex and revitalization of the tooth as well as replacement of lost dentin by newly formed dentin should be ultimate objectives of these treatment strategies.

Caries is a biofilm mediated disease of the hard tissues of teeth that is caused by bacterial conversion of fermentable carbohydrates into acids resulting in a acidogenic and cariogenic environment which eventually breaks down the dental hard tissues to form a cavity.

Caries of the permanent teeth was reportedly the most common oral condition as per the Global Burden of Disease Study of 2017. Globally, around 2.4 billion people suffer from caries of the permanent teeth and 486 million children suffer from caries of the primary teeth. The overall prevalence for Dental caries in India is about 54.16%. However there is a remarkable variation in dental caries prevalence rates as per age, diagnostic criteria, dentition, and geographical region.

Involvement of the dentin-pulp complex in the carious process is associated with an inflammatory response. The histopathology and the pathophysiology of the diseased pulp have been extensively studied in the literature clearly illustrating that the parts of the pulpal organ under the inflamed pulpal tissue even in so called "irreversible pulpitis" remain vital or if slightly inflamed are often capable of retaining their vitality especially in the radicular portion. Therefore, there is a growing focus on conserving pulp vitality in different types of teeth with pulp involvement.

Vital pulp therapies are a collection of treatment procedures that aim to conserve the vitality of the pulpal tissue that is affected by the carious process. The procedures include removing the microbial irritation and preventing any new bacterial insult to the pulp by placement of a sealing biocompatible material to protect the pulp from external stimuli. VPT is easier and less invasive than conventional root canal treatment. However the technique is still demanding often requiring magnification and expertise.

Vital pulp therapies have become common in recent years also in part due to the development of highly biocompatible materials like MTA and various formulations of calcium silicate based materials. Calcium hydroxide based pulp therapies have nearly been replaced by MTA; MTA and calcium silicates are now recognized as the benchmark for vital pulp therapies.

A procedure termed 'miniature pulpotomy' has been proposed to improve outcomes of direct pulp capping. By removing the superficial pulp (about 1mm) under a deep carious lesion on a tooth with reversible pulpitis, infected dentin chips and inflamed pulp might be removed to give better access to highly biocompatible materials (MTA and calcium-silicate based materials) as well as provide a clean surgical wound for repair.

The ESE (European Society of Endodontology) and the AAE (American Association of Endodontists) have conflicting guidelines regarding the management of deep and extremely deep carious lesions. The ESE defines Deep caries as 'Caries reaching the inner quarter of dentine, but with a zone of hard or firm dentine between the caries and the pulp, which is radiographically detectable when located on an interproximal or occlusal surface having risk of pulp exposure during operative treatment'.

On the other hand, extremely deep caries is defined as Caries penetrating the entire thickness of the dentine, radiographically detectable when located on an interproximal or occlusal surface. Pulp exposure is unavoidable during operative treatment. The ESE position statement recommends 'Selective caries removal' whereas the AAE recommends complete caries excavation to eliminate the infection in its totality. The Indian Endodontic society (IES) considers VPT as the 'cornerstone of modern endodontics' in management of deep carious lesions and exposed pulps.

By delving into the realm of regenerative dentistry, the exploration of regenerating dental tissues through the art of tissue engineering has stood as a fervent focus of recent research. Structures resembling teeth have successfully been cultured in laboratory environments. Regeneration of dentin has been the most relevant and accessible form of tissue engineering since the dentin forming cells- the odontoblasts stay functional throughout the life of the vital tooth. Tissue engineering (TE) is a branch of regenerative medicine that combines materials science, applied cell biology, and medical engineering to replace or restore organ function. The prevailing technique in tissue engineering involves seeding cells into scaffolds. These are three-dimensional structures that serve as an extracellular matrix, creating a conducive environment for cell growth and development. Ideally, a scaffold should possess the following attributes: an appropriate surface for cell attachment, porosity and permeability to facilitate cell movement and nutrient penetration, and ultimately degrade into harmless and benign compounds. An optimal scaffold may also be shaped to direct cell adhesion, proliferation, migration, and spatial organization since scaffolds provide the blueprint for these processes.

Scaffolds, stem cells, and growth factors form the fundamental components for the regeneration of any tissue. Diverse scaffolds have been researched for dentin regeneration, encompassing synthetically-engineered polymeric and ceramic scaffolds such as synthetic polymers (PLA, PGA, PLGA) as well as naturally derived options like collagen, chitosan, cellulose, alginate, gelatin, among others.

Recently, Treated dentin matrix, an extracellular matrix-based biomaterial, has emerged as an excellent scaffold for tissue engineering because of its remarkable biological induction activity, distinct natural structure, and biocompatibility. In addition to having a high level of bioactivity, a treated dentin matrix can work as a transporter for bioactive substances and medication molecules, aiding in the processes of tissue regeneration and immunomodulation. Similar products such as demineralized bone matrices (DBMs) and other allograft bone materials have already found their place in clinical practice.

Comparative evaluation of calcium silicate-doped treated dentin matrix and mineral trioxide aggregate as miniature pulpotomy biomaterials in deep carious lesions: a parallel, double-blind, randomized clinical trial.

AIM:

To compare the efficacy of a Novel calcium silicate doped treated dentin matrix and Mineral Trioxide aggregate as biomaterials for miniature pulpotomy.

OBJECTIVES:

Primary objective:

To evaluate the efficacy of calcium silicate-doped human-treated dentin matrix (CaSi+hTDM) compared to Mineral Trioxide Aggregate (MTA) in maintaining pulp vitality using cold testing following Miniature Pulpotomy (MP) in deep and extremely deep carious lesions with reversible pulpitis in 14- to 35-year-old patients reporting to Department of Dentistry, AIIMS Nagpur.

Secondary objectives:

1. To evaluate patient-reported outcomes such as pain, swelling, sinus tract etc. post-operatively.
2. To determine the clinical success rates of both materials by assessing the Periapical index of healing over a 6 months follow-up period.

NULL HYPOTHESIS:

The null hypothesis (H0) is that there is no difference between CaSi+hTDM and MTA in maintaining pulp vitality when used as a Miniature Pulpotomy (MP) biomaterial in carious lesions.

Literature Review:

Vital pulp therapy is defined as a treatment aimed at conserving and sustaining compromised dental pulp tissue that has been impacted by extensive dental caries, dental trauma, and restorative interventions. or due to other iatrogenic reasons. Pulp preservation and vital pulp therapies have taken center stage in the last few years. It is important to take into consideration the entire history and genesis of pulp preservation techniques along with the newer ones that are becoming popular. Pulp preservation techniques are quite old, with reports of gold being placed directly over the injured pulp by Pfaff in the 18th century. In the early nineteenth century, the concept of pulp capping primarily revolved around the belief that pulpal healing took place solely following the etching and cauterization of the pulp. Numerous breakthroughs in the realms of medicine and technology, such as the discovery of microorganisms by Robert Hooke and Antoni van Leeuwenhoek, role of microorganisms in pathogenesis of various diseases by Pasteur and Lister, the introduction of dental radiographs in 1895 and development of anesthesia by Horace Wells and Willian Morton, has tremendously helped shape our understanding of the physiology of the pulp as well as pathology and treatment of pulpal and periapical diseases. The first clinical scientific study comparing different pulp capping materials done by Dätwyler demonstrated that zinc oxide eugenol showed the best results. After the introduction of Calcium hydroxide by Herman in 1920, numerous studies were conducted, indicating its biocompatibility when applied over vital pulp. Despite the perception in the early 1900s that an exposed pulp was deemed a 'doomed organ', it was not until research investigating pulp healing and pulpal responses to injuries and pulp capping materials were carried out, which helped in elevating our understanding of the injured pulp while also showing the unpredictability of outcomes for direct pulp capping. Success rates at that time were about 60-70% for direct pulp capping compared with 80-90% for RCT. Vital pulp treatments using calcium hydroxide had several drawbacks, such as inadequate adherence to dentin, gradual dissolution over time, and microleakage issues. However, with the introduction of Calcium silicate cements and improvement of our understanding of pulpal repair, there has been a profound change in our perspective regarding vital pulp therapies and hence this has translated to good clinical results for pulp capping and pulpotomy. Numerous great reviews have been done on the subject of Vital pulp therapies and their future directions.

Newer Definitions of VPT have been simplified to include all; 'Strategies aimed at maintaining the vitality of the pulp'. This includes one- and two-step selective caries removal techniques and indirect pulp capping to avoid pulp exposure as well as direct pulp capping and pulpotomy procedures. Recent position statements from the AAE and the ESE have provided conflicting recommendations for VPT's. The ESE position statement recommends 'selective carious-tissue removal (one-stage or two-stage stepwise technique) in teeth with reversible pulpitis, provided radiographic assessment indicates caries has progressed no deeper than the pulpal quarter with a zone of dentin separating the carious lesion from the pulp chamber'. On the contrary, the AAE recommends that 'complete caries removal is essential to eliminate infected tissues and visualize pulp tissue conditions under magnification when pulpal exposures occur. Residual caries compromises necessary observations of pulpal inflammation levels for a diagnosis of more severe pulpitis'. In instances when pulpitis was more severe, the ESE recommended that 'carious exposure with symptoms indicative of irreversible pulpitis should be treated aseptically with pulpectomy. Alternatively, full pulpotomy may be successful in cases where there is partial irreversible pulpitis in the coronal pulp; however, better long-term prospective randomized data are required'. The AAE have limited their recommendations to 'utilizing direct visualization of the pulp, it appears that even symptomatic pulps may be candidates for VPT'. Hence due to the conflicting recommendation, ways to improve the decision-making process is of paramount importance to improve the consistency and predictability of VPT. In management of deep carious lesions, carious exposures with signs and symptoms indicative of irreversible pulpitis, removal of pulp tissue either in a partial pulpotomy or full pulpotomy since the carious lesion has progressed into the pulp and there is bacterial infiltration along with concomitant pathological alterations in the pulp. Recently development of inflammatory and other biomarkers which accurately reflect the level of inflammation in the pulp offer objective means of measuring pulp inflammation. However, this requires exposure of pulp since volume retrieved from dentinal fluid in unexposed cavities is likely to be too small for analysis.

For pulp capping, calcium hydroxide was regarded for many years as the gold standard because of its potent antibacterial properties. However disadvantages included inflammation of pulpal surface and necrosis, formation of tunnel defects in newly formed dentin, high solubility in oral fluids and lack of adhesion.

MTA (Mineral Trioxide Aggregate) was first introduced in the 1990s as an experimental calcium silicate-based material. Its composition primarily comprises Portland cement, which contains tricalcium and dicalcium silicate, along with bismuth oxide serving as a radiopacifier. Commercial forms of MTA include ProRoot® MTA and tooth coloured ProRoot® MTA, (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA), and MTA Angelus® and MTA Bianco®, (Angelus, Londrina, Brazil). MTA has a variety of uses in Endodontics including being the material of choice in cases of pulp capping, pulpotomies, perforative root resorption defects, surgical root end filling, root and pulp chamber perforations and in revascularization cases MTA has demonstrated both inductive and conductive properties for promoting hard tissue formation. It also stimulates the formation of cementum-like hard tissue and contributes to bone regeneration. A randomized controlled trial, concluded that MTA exhibited greater clinical ease of use, led to reduced pulpal inflammation, and yielded more predictable outcomes for hard tissue barrier formation in comparison to calcium hydroxide for pulp capping procedures. In a meta-analysis, it was demonstrated that MTA had significantly higher success rates compared to calcium hydroxide (CH). MTA specimens exhibited lower levels of pulpal inflammation than CH specimens and showed a higher percentage of calcified dentin bridge formation as well. Despite its numerous advantages, MTA does have some drawbacks, such as challenges in handling, a prolonged setting time, higher cost, and the possibility of tooth discoloration. Biodentine (BD), developed by Septodont, France, is a calcium silicate-based Portland cement. It finds application in direct posterior restorations, addressing furcal perforations, performing retrograde filling, and for pulp capping procedures. Biodentine is regarded as a viable alternative to MTA due to its superior mechanical properties and favorable handling characteristics.

Recently, Bioceramics have been introduced like the IRoot BP Plus (Innovative Bioceramix, Vancouver, Canada) also labelled as EndoSequence Root Repair Material Putty (ERRM) (Brasseler, Savannah, GA, USA) and as TotalFill RRM Putty (FKG, La-Chaux-de-Fonds, Switzerland). The main composition of these materials being tri-calcium silicate, bi-calcium silicate and calcium phosphate. iRoot BP plus has good biocompatibility with the pulp tissue and induced formation of a reparative dentin bridge, it therefore can be used as a pulp capping material.

Various criteria are used to define the success of Vital pulp therapies in the literature. Maintenance of pulpal health both clinically and radiographically, dentin deposition over the material placed close to the pulp, absence of postoperative pain and discomfort are some of success defining criteria present in the literature.

One of the primary objectives of the vital pulp therapy is to encourage formation of a protective hard tissue barrier after an injury. The process of forming a hard tissue barrier begins with the recruitment of odontoblast-like cells from the cell-rich zone and sub-odontoblastic layer, which leads to tertiary dentin deposition under the material.

Even though currently available calcium silicate based materials support mineralization and cell growth, they are not able to provide a signal for odontogenic differentiation as well as dentin regeneration. Due to the limitations of these materials naturally derived materials have been tried. Hence, to provide a better strategy for dentin regeneration, tissue engineering concepts have been introduced for vital pulp therapies.

Scaffolds are an important part of tissue engineering. The goal of tissue engineering is to create a three-dimensional complex of biomaterials and cells that resembles biological tissue. This complex can then be utilised to replace the injured organ permanently by reconstructing its appearance, structure, and function. The triad of tissue engineering consists of a scaffold, stem cells and growth factors. Scaffolds used for dentin and pulp tissue regeneration encompass a range of materials. Natural scaffolds include collagen, glycosaminoglycan, chitosan, alginate, and agarose. Synthetic options comprise hydroxyapatite/tricalcium phosphate, polyacetic acid, polycaprolactone, and self-assembling peptide hydrogels.

Research on polysaccharide-based scaffolds like alginate scaffolds has revealed that Human Dental Pulp Cells (HDPCs) can effectively differentiate into odontoblast-like cells and stimulate calcification processes that closely mimic dentin formation. These findings support the use of alginate as a promising scaffold for dental tissue regeneration. Alginate offers several advantages, including its biocompatibility and non-immunogenic nature. However, it has disadvantages such as poor cell adhesion, low mechanical strength, and limited degradability. Chitosan is naturally found in the exoskeletons of marine crustaceans like shrimps and crabs, as well as in the cell walls of fungi. There have been conflicting findings regarding chitosan as a scaffold. While some studies have shown that a 3D chitosan scaffold supports the differentiation of Dental Pulp Stem Cells (DPSCs) due to its suitability for nerve cell attachment, other studies may have reported different outcomes or challenges with chitosan scaffolds in certain applications. But The results from Kim et al. indicated that when chitosan was compared to other natural scaffolds such as collagen and gelatin, these latter materials better supported the growth of Human Dental Pulp Cells (HDPCs). Due to its poor solubility chitosan has to be modified in order to be utilized in regenerative dentistry.

Extracellular matrix based scaffolds like hyaluronic acid is a linear polysaccharide abundant in cartilage ECM. Because of its high molecular weight, when dissolved in water, its viscoelasticity increases making it easier to be used as an injectable scaffold. Advantages include its bioactivity, biocompatibility, biodegradability and ability to act as a growth factor reservoir; disadvantages however include structural complexity, low mechanical strength and possible immunogenicity. Collagen is one of the most abundant components of extracellular matrices. Most abundant types of collagen used in tissue engineering is collagen type I and allogenic collagen such as bovine collagen which has great biocompatibility and bioactivity. Advantages of collagen include its great mechanical properties and ability of collagen to induce DPSCs into highly vascularized and organized matrix of odontoblast like cells.

Scaffolds derived from proteins include Fibrin based scaffolds like Platelet-rich fibrin (PRF) which is considered as a second generation platelet concentrate, is known to be rich in platelets, leukocytes and numerous growth factors that play an important and essential role in promoting cell proliferation and differentiation. PRF acts as a 3D mesh that can capture migrating cells and induces release of platelet derived growth factors. PRF has been tested as a pulp capping material in canines and it shows promising results for regeneration of pulp as it supplies numerous growth factors. A study compared different types of scaffolds for inducing apexogenesis in necrotic immature permanent teeth. Within the four scaffolds used, blood clot, PRF, collagen and PLGA; PRF exhibited the best results for all testing parameters. Peptides are short amino acids sequences of proteins that have biological properties. Peptides are highly customizable in regards to their biological, physical and chemical properties. Self-assembling peptides are modified peptide molecules that are self-assembled into fibrillary structures and offer advantages in regenerative endodontics like mimicking the extracellular matrix due to its nanoscale dimensions.

Growth factors(GF) are groups of proteins which bind to cell receptors and induce cellular proliferation and differentiation. It also refers to the extracellular signals that control organogenesis and morphogenesis during interactions between mesenchymal and epithelial cells. Growth factors are one of the main components of tissue engineering or any regenerative procedure. They are key factors for tissue wound healing by regulation of immune function, proliferation and differentiation of cells. Several growth factors are potential therapeutic agents for hard tissue regeneration. Some are used to increase stem cell numbers such as the platelet derived growth factors (PDGF), fibroblasts growth factors (FGF), colony stimulating factors (CSF) and epidermal growth factors (EGF). Others modulate and control humoral and cellular responses such as Interleukin-12 and Insulin-like Growth Factor 1 (IGF1) especially in activation and survival of antigen specific T cells. Dentin matrix also releases various proteins like TGF Beta-1, COL-1, DMP-1, decorin and DSP which have been found to stimulate dentinogenesis.

For pulp capping materials scaffolds can thus be mixed with growth factors and this has shown superior results enhancing reparative dentinogenesis. In a study, odontoblast-like cellular differentiation and upregulation of matrix secretion in human dentin pulp complex was shown when TGF-Beta 1 was incorporated in alginate hydrogel scaffold. When comparing the effects of MTA alone versus MTA combined with fibroblast growth factor-2 (FGF-2) in vitro on human dental pulp cell behavior, the study concluded that the MTA and FGF-2 group significantly enhanced human dental pulp cell proliferation and promoted osteogenic differentiation. Furthermore, the combination of both MTA and growth hormone (GH) was found to promote cell adhesion, growth, differentiation, and angiogenesis by activating bone morphogenetic proteins and the Mitogen-Activated Protein Kinase (MAPK) pathway.

A treated dentin matrix (TDM) is a special kind of decellularized extracellular matrix (dECM) that originates from dentin matrix (DM). A Scaffold derived from dentin is the best option we have for achieving the ideal imitation of dentin tissue. As a result, TDM has been extensively studied in recent years. TDM preserves the basic structure of natural dentinal tubules, allowing stem cells to adhere and provide the necessary space for nutrient and metabolic waste exchange. It also exposes various and abundant bio-active proteins, such as growth factors, to better induce stem cell proliferation, adhesion, and differentiation to promote dental pulp, dentin, cementum, periodontal ligament, and alveolar bone regeneration. Furthermore, TDM is able to serve as a carrier and release controller for some drug molecules and bio-active agents by taking advantage of its unique structure of exposed dentinal tubules.

In the literature several techniques have been tried for fabrication of treated dentin matrix. The essential steps in the fabrication approach for TDM are typically as follows: extraction of teeth, removal of enamel, cementum and dental pulp, sectioning into matrixes or pulverization into particles, demineralization, specific treatment (if required), sterilization, and preservation. One study detailed the different fabrication and preservation techniques. Extracted human teeth are the most common source for harvesting TDM. Studies using animal TDMs, including goats, canines, monkeys, and pigs, demonstrate that these are also feasible. It is important to remember that pig TDM and human TDM have comparable mineral phases, bioactive compounds, and odontogenic induction abilities.

In addition to this, several investigators have used special treatments on TDM and obtained various results. Studies have shown that Atelopeptidization of demineralized dentin could facilitate preserving the collagen structure and reducing the immune reaction. Another study used ethanol/DMA solution and showed that it might be capable of enhancing the mechanical properties of demineralized dentin matrix. Another study freeze dried the dentin matrix and showed that freeze-dried dentin matrix has similar mechanical and biological properties of those of dentin.

One study showed that both human dentin particulates and deproteinized bovine bone matrix supported cell proliferation in DPSCs. Another study showed a Dose-dependent promotion of cell proliferation with a higher concentration of the dentin matrix components on OD-21 cells. A treated dentin matrix paste significantly promoted cell proliferation in DPSCs in another study. However, in a different study by, treated dentin matrix extracts combined with dental pulp-cell derived small extracellular vesicles suppressed cell proliferation. Another study showed that mRNA expressions of OCN, DSPP, VEGF-1 and Nestin was upregulated by a hTDM leaching solution. Another significant study showed that TDM paste significantly enhanced the expressions of ALP, BSP and DSP in DPSCs. TDM has the capacity to cause mesenchymal stem cells to develop into osteoblasts and odontoblasts. Induced mesenchymal cells expressed more odontogenic and osteogenic-related genes and proteins.

Dental pulp stem cells (DPSCs), dental follicle cells (DFCs), cranial neural crest cells(CNCCs), umbilical cord mesenchymal stem cells(UCMSCs) and bone marrow stromal cells(BMSCs) were employed to explore the effect of a treated dentin matrix on cell differentiation by means of polymerase chain reaction, Western blot assay or immunostaining. Induction of both DFCs and DPCs by treated dentin matrix to display odontogenic differentiation potential was shown in a study.

A study has shown that new dentin was formed in a rat mandible cultured with a treated dentin matrix and DPSCs. While another showed that TDM induced DPSCs to regenerate dentin-like tissues expressing DSPP and DMP-1. Another study by the same author on DFCs showed that hTDM induced complete dentin tissue regeneration that expressed DSP and DMP-1. In a different study, the author developed a treated dentin matrix hydrogel (TDMH) for direct pulp capping, which played a role in achieving dentin regeneration while also preserving pulp vitality. CBCT showed TDMH-induced superior dentin bridge formation of higher radiodensity and thickness than Biodentine and MTA. Histological analysis showed TDMH induced thicker dentin with layers of well-arranged odontoblasts than Biodentine and MTA. In a study, it was demonstrated that Treated Dentin Matrix Paste (TDMP) stimulated the formation of a continuous reparative dentin bridge that was thicker and denser compared to calcium hydroxide. TDMP achieved both dentin regeneration and vital pulp conservation.

In conclusion, TDM is a versatile biomaterial application of which will not be restricted to the field of just dental research. Thanks to the unique porous structure and growth factors preserved within, TDM exhibits the ability to contribute to bone regeneration, soft-hard tissue interface reconstruction and immunomodulation with its own endogenous bio-active molecules and carried exogenous drugs.

Recently Calcium-silicate based materials like calcium-enriched mixture (CEM) and Biodentine have been used widely for Vital pulp therapy. CEM cement has similar physical properties to MTA and has shown PDL regeneration, cementogenesis and dentinogenesis in animal studies. It is also capable of stimulating dentinal bridge formation. Biodentine is another calcium-silicate based material that also provides complete dentinal bridge formation with absence of an inflammatory response. Calcium silicate-based materials have been demonstrated to support dental pulp stem cell proliferation and growth, while also upregulating the expression of genes such as DSPP (Dentin Sialophosphoprotein) and DMP1 (Dentin Matrix Protein 1). Hence calcium silicate is a great biocompatible material for vital pulp therapy.

The literature is scarce regarding miniature pulpotomy procedure. Only a few case reports have been published regarding this procedure, demonstrating its applicability in treating symptomatic mature molars diagnosed with irreversible pulpitis.Only a single randomized clinical trial has been done using this procedure.

MATERIALS AND METHODS:

Study Design:

This will be a prospective, block-randomized, double-blinded, and parallel-group clinical trial. The study will obtain ethical clearance from the Institutional Ethics Committee, and the protocol will be registered in the Clinical Trial Registry of India, ensuring adherence to ethical standards and transparency in research procedures. All the procedures will be followed conforming to the Helsinki Declaration of the World Medical Association. A patient information sheet and consent form will be distributed to all participants.

Study Setting:

AIIMS Nagpur is a premier medical institution in India, known for its advanced medical care, research, and education. It is located in MIHAN, Nagpur, Maharashtra. It is easily accessible via major transport links, making it convenient for participants to attend follow-up visits. The Dentistry OPD at AIIMS Nagpur serves a large number of patients daily, providing ample recruitment opportunities for study participants. It is equipped with modern dental chairs, advanced diagnostic tools (such as digital radiography), and treatment facilities. A robust electronic medical records (EMR) system ensures accurate data collection and management, facilitating longitudinal follow-up of patients. The cost of treatments available in AIIMS is affordable and minimal when compared to other hospitals and private clinics.

Clinical Setting

Treatment rooms are equipped with dental chairs and necessary

ELIGIBILITY:
Inclusion Criteria:

* The healthy participants (ASA 1 and 2), between ages 14 - 35 years, reporting to AIIMS Nagpur from within a 100 kms radius with carious pulp exposure in mature permanent teeth and with the following clinical and radiographic features will be included in the study:

I. Clinical features

1. The clinical diagnosis of reversible pulpitis characterized by mild pain (on Numerical Rating Scale 11) that goes away within a couple of seconds following the removal of the stimulus (113)
2. Positive response to pulp sensibility tests.

II. Radiographic features

1. Normal periapical tissues [Periapical index (PAI) score ≤2](114)
2. The presence of carious lesion with radiolucency penetrating three-fourths (deep caries) or the entire (extremely deep caries) dentin thickness

Exclusion Criteria:

* The patients with the following clinical and radiographic features will be excluded from the study:

I. Clinical features

1. A history of spontaneous unprovoked toothache, pain on percussion, a sinus tract, compromised periodontal status (periodontal pockets > 4mm), excessive mobility, crack
2. Profuse hemorrhage from exposure site (>5 minutes)
3. The presence of serous or purulent exudates from the exposure site.
4. Teeth that have experienced traumatic occlusion, non-carious lesions, developmental defects etc.

II. Radiographic features

1. The evidence of internal or external resorption, or the calcification of the pulp chamber or canals or presence of condensing osteitis.
2. The presence of radiolucency in the furcation or periapical regions.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pulp vitality | From enrollment to the end of treatment at 6 months
  Pulp vitality assessed by cold testing

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS Nagpur, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clementino MA, Gomes MC, Pinto-Sarmento TC, Martins CC, Granville-Garcia AF, Paiva SM. Perceived Impact of Dental Pain on the Quality of Life of Preschool Children and Their Families. PLoS One. 2015 Jun 19;10(6):e0130602. doi: 10.1371/journal.pone.0130602. eCollection 2015. PMID 26090927